CLINICAL TRIAL: NCT02899429
Title: Systematic Descriptive Experimental Ultrasound Study of Entheses and Small Joints of Hands and Feet in Patients Presenting an Atypical Form of Psoriasis
Brief Title: Ultrasound Study of Entheses and Small Joints of Hands and Feet in Patients With Atypical Form of Psoriasis
Acronym: ECHOPSO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ECHOPSO (RB14.120)
Record Dates: First submitted 2016-08-30; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Ultrasound in Patients With Atypical Shape of Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Systematic study of the ultrasound infringements of tendons chest expanders of entheses the most involved in spondylarthropathies and small joints of hands and feet in expanding patients of psoriasis to estimate if there is an infra-clinical infringement of the psoriasic rheumatism .

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Atypical psoriasis of the scalp and / or nails and / or psoriasis of folds
* Patient agreeing to participate in the study

Exclusion Criteria:

* Psoriatic arthritis
* Rheumatic pain
* Arthritis
* Joint Trauma in hands, elbows knees, feet
* Current treatment with methotrexate, soriatane, cyclosporine, corticosteroids
* Current treatment with biological therapy (anti-TNF, anti IL 12-23)
* Previous history of rheumatic disease: inflammatory, microcrystalline, osteoarthritis
* Patients in physical or mental incapacity to agree

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient with atypical cutaneous psoriasis consultant at University Hospital of Brest
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Infra clinical infringements of the entheses | 1 year
  Measurement of the thickness in millimeters (mm) in anteroposterior diameter of each entheses (quadricipatal tendon, calcaneal tendon and plantar aponeurosis)
Infra clinical infringements of the nails | 1 year
  Measurement mm of the nail plate and matrix of the nail. It will be evaluate by using power Doppler the vascularisation in 3 grades of the nail ( grade 0=normal, grade 1=moderate vascularisation , grade 3:= abnormal vascularisation)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Jousse, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France